CLINICAL TRIAL: NCT02129127
Title: First in Human Evaluation of the Drug-Coated Chocolate Balloon for Percutaneous Transluminal Revascularization of Infrainguinal Arterial Disease
Brief Title: Drug-Coated Chocolate PTA Balloon in Patients With Peripheral Arterial Disease - The ENDURE Trial
Acronym: ENDURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriReme Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP004
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug Coated Chocolate (Experimental): Paclitaxel Coated Chocolate Balloon Angioplasty
  Interventions: Device: Paclitaxel Coated Chocolate Balloon Angioplasty

INTERVENTIONS:
Device: Paclitaxel Coated Chocolate Balloon Angioplasty — Balloon Angioplasty with the Chocolate Balloon resulting in vessel dilatation and localized delivery of Paclitaxel

SUMMARY:
This first-in-man study is to evaluate the Drug-Coated Chocolate (DCC) Balloon for percutaneous arterial angioplasty in patients with symptomatic peripheral arterial disease. The study focuses on acute device performance and peri-procedural safety and also seeks to further characterize the performance of the device.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm study. Symptomatic lower extremity Peripheral Arterial Disease (PAD) patients presenting for endovascular revascularization will be enrolled in the study if they meet all entry criteria. The study will include patients from New Zealand and the European Union. The endpoints were designed to establish safety of the DCC and to identify long-term clinical benefits of this technology.

The patients treated in this study will be designated into the above the knee (ATK) follow-up schedule if they are treated with the DCC in the SFA or Popliteal vessels. This schedule calls for clinical visits with duplex ultrasounds at 1,6 and 12 months. Patients will be designated into the below the knee (BTK) follow-up schedule if they are treated with the DCC in the Peroneal, Anterior Tibial, Posterior Tibial or Pedal vessels. These patients will have clinical visits at 1, 3 and 6 months with duplex ultrasound at the 1 and 6 months visits only.

ELIGIBILITY:
Key Inclusion Criteria:

* Intermittent claudication or critical limb ischemia
* Atherosclerotic target lesion >70% stenosis
* Reference vessel diameter (RVD) between 2.0 and 6.0mm
* Angiographic evidence of distal run-off
* Target lesion length <150mm that consists of no more than two adjacent lesions( < 25mm apart) and is able to be completely covered with inflation of no more than two DCC devices

Key Exclusion Criteria:

* Acute limb ischemia or thrombolytic therapy
* Known and relevant allergies/hypersensitivities
* Known impaired renal function
* Known bleeding disorder
* Severe calcification at the target lesion
* Previous bypass or stent at, or proximal to, target vessel
* Aneurysm in target limb
* Prior major limb amputation
* Use of a any of the following: re-entry device, atherectomy, laser or other ablation procedure, or cutting/scoring balloon at the target lesion; use of drug eluting stent, or non-study drug coated balloon in the target limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Late Lumen Loss (LLL) | 3 Months (BTK) or 6 Months (ATK)
  LLL is determined by assessing the difference between the minimum lumen diameter (MLD) immediately after treatment with the DCC and the MLD at angiographic follow-up. LLL will determined by the Angiographic Core Laboratory.

SECONDARY OUTCOMES:
Device Success | approx 1 hour
  This is defined as the percentage of procedures that accomplish less than 30% residual stenosis without flow-limiting dissection at target lesion after DCC treatment.
Technical Success | approx 1 hour
  This is defined as the percentage of cases in which the DCC is able to be delivered to and inflated at the intended target lesion location successfully.
Device Related Adverse Events (AEs) | 30 days
  Occurrence and Severity of any DCC Related AEs will be analyzed
Freedom from Target Lesion Revascularization (TLR) | 30 days / 3 Months (BTK only) / 6 Months / 12 Months (ATK only)
  This will calculate the number of patients who do not require a clinically indicated TLR. Clinically indicated TLR is defined as any repeat percutaneous intervention at the DCC target lesion or bypass surgery at the DCC target vessel performed for >50% restenosis or another complication of the target lesion
Amputation Free Survival | 30 days / 3 Months (BTK only) / 6 Months / 12 Months (ATK only)
  This is a composite endpoint which counts the number of patients who experience limb salvage. Patients will fail this endpoint if they undergo a major amputation (defined as unplanned amputation at or above the ankle) or if a procedure related death occurs.
Patency | 6 Months / 12 Months (ATK only)
  The percentage of cases in which the treated lesion is patent. Patency is demonstrated by a Peak Systolic Velocity ratio <2.5 at the target lesion assessed on Duplex Ultrasound without the need for re-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, MD, Principal Investigator — Auckland City Hospital; Thomas Zeller, MD, Principal Investigator — Universitats Herzzentrum Bad Krozingen
Locations (2):
- Universitats Herzzentrum Bad Krozingen, Bad Krozingen, Germany
- Auckland City Hospital, Auckland, New Zealand